CLINICAL TRIAL: NCT03088527
Title: A Phase 1, First-in-Human, Multi-Part Study of RAD140 in Postmenopausal Women With Hormone Receptor Positive Breast Cancer
Brief Title: Phase 1, First-in-Human Study of RAD140 in Postmenopausal Women With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD140-01-001
Record Dates: First submitted 2017-02-28; First posted 2017-03-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast
MeSH Terms: interventions — RAD140

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAD140 Part A and Part B (Experimental): Part A, Dose Escalation: Patients will be assigned sequentially to escalating doses of RAD140.
  Part B, Safety Expansion: Once the maximum tolerated dose (MTD) has been identified and/or a recommended dose escalation (RDE) has been determined, additional patients will be enrolled to further evaluate the safety, tolerability and preliminary clinical activity of the recommended dose.
  Interventions: Drug: RAD140

INTERVENTIONS:
Drug: RAD140 — RAD140 will be supplied as formulated drug-in-capsules for oral administration.

SUMMARY:
The primary purpose of this study is to evaluate the clinical safety profile, tolerability, and pharmacokinetic (PK) characteristics of RAD140 in hormone receptor positive breast cancer.

DETAILED DESCRIPTION:
This is a first in humans study that is designed to evaluate the clinical safety profile, tolerability, and pharmacokinetic (PK) characteristics of RAD140 in hormone receptor positive breast cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Progressive metastatic or locally advanced or metastatic breast cancer.
* Clinically confirmed as postmenopausal.
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 1 at screening.

Key Exclusion Criteria:

* HER2 positive patients by local laboratory testing.
* Triple negative breast cancer.
* Any chemotherapy within the 28 days prior to the first dose of study drug.
* Any non-chemotherapy anti-cancer drug less than 5 half-lives (30 days for biologics) or less than 14 days for small molecule therapeutics, or if half-life is not known.
* Tamoxifen and aromatase inhibitors within 14 days prior to the first dose of study drug.
* Fulvestrant within 30 days prior to first dose of study drug.
* Any investigational drug therapy within 5 half-lives of the previous investigational study drug or 30 days, whichever is shorter.
* Radiation therapy for breast cancer within 2 weeks of dosing and planning to have radiation therapy during participation in this study.
* Known history of human immunodeficiency virus infection (HIV) or hepatitis C or active hepatitis B infection, unless the patient was diagnosed >10 years prior to enrollment and no evidence of active liver disease.
* Currently taking testosterone, methyltestosterone, oxandrolone (Oxandrin), oxymetholone, danazol, fluoxymesterone (Halotestin), or testosterone-like agents.
* Untreated or uncontrolled brain metastasis.
* Diagnosed with or treated for cancer within the previous 2 years, other than breast cancer or non-melanoma carcinoma of the skin.
* Pregnant and nursing females.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose-limiting toxicities (DLTs) RAD140 treatment | First 28 days of treatment
  Incidence rate of dose-limiting toxicities (DLTs) RAD140 treatment
Number of adverse events related to study treatment | Up to 30 days after end of treatment
  Number of adverse events related to study treatment
Number participants with dose interruptions and dose adjustments | Up to 30 days after end of treatment
  Number participants with dose interruptions and dose adjustments

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 1 and 15
  Maximum plasma concentration (Cmax)
Time to maximum plasma concentration (Tmax) | Day 1 and 15
  Time to maximum plasma concentration (Tmax)
Area under the plasma concentration versus time curve (AUC) | Day 1 and Day 15
  Area under the plasma concentration versus time curve (AUC)
Tumor response | Screening and every 8 weeks for up to 12 months of treatment
  Clinical benefit rate (CBR) or objective response rate (ORR) will be assessed by Investigators per RECIST v1.1 along with time-related efficacy endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Clinical Operations, Study Director — Radius
Locations (5):
- United States (5):
  - Yale Cancer Center, New Haven, Connecticut
  - Cancer Center Protocol Office, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No